CLINICAL TRIAL: NCT00767052
Title: A Randomised Single Centre Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetics of Oral Multiple Ascending Daily Doses of AZD1236 Tablet by a Single-Blind, Placebo-Controlled, and Single Dose Relative Bioavailability of the Oral Suspension and Oral Tablet Formulations by an Open Cross-Over in Healthy Japanese Men
Brief Title: Investigate the Safety Tolerability and Pharmacokinetics of Multiple Doses of AZD1236
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: J Andrew Lockton MRCP(UK) MD FFPM, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D4260C00006
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Safety; Tolerability; Pharmacokinetics; AZD1236
MeSH Terms: interventions — 4-((5-chloro-2-pyridinyl)oxy)-1-((((4S)-4-methyl-2,5-dioxo-4-imidazolidinyl)methyl)sulfonyl)-piperidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active (Experimental): AZD1236 tablet
  Interventions: Drug: AZD1236
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo
- Relative bioavailability (Other): AZD1236 Oral suspension
  Interventions: Drug: AZD1236
- Relative bioavailability tablet (Other): AZD1236 tablet
  Interventions: Drug: AZD1236

INTERVENTIONS:
Drug: AZD1236 — 75mg once daily or 75mg twice daily will be administered in multiple dose part.
  Arms: Active
Drug: Placebo — Placebo tablet matching to the active in multiple dose part.
  Arms: Placebo
Drug: AZD1236 — 75mg single dose will be administered in relative bioavailability part.
  Arms: Relative bioavailability
Drug: AZD1236 — 75mg oral suspension single dose will be administered in relative bioavailability part.
  Arms: Relative bioavailability tablet

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of multiple ascending oral doses of AZD1236 given to healthy young subjects for 13 days and to evaluate the single-dose relative bioavailability of the oral suspension and oral tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Body Mass Index (BMI) between 19-27 kg/m2

Exclusion Criteria:

* Receipt of another investigational drug in the 4 months before dosing in this study
* Acute illness which requires medical intervention within 2 weeks of Visit 2.
* Abnormal resting BP and pulse rate (after resting for 10 minutes). Supine blood pressure > 140 mmHg systolic or >90 mmHg diastolic, pulse<= 50 or => 90 beats per minute

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD1236 by assessment of blood pressure, pulse rate, body temperature, laboratory variables, ECG and adverse events | Assessments taken at screening visit, defined timepoints pre-dose and post-dose during treatment periods and follow up visit. Volunteers will be monitored throughout the study for adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD1236 in blood | Samples taken during Visit 2 in multiple dosing part at 41 points and Visit 2/3 in relative bioavailability part at 32 points.

CONTACTS AND LOCATIONS:
Overall Officials: Shunji Matsuki, MD PhD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Osaka, Osaka, Japan